CLINICAL TRIAL: NCT04171635
Title: Quantitative Susceptibility Mapping (QSM) to Guide Iron Chelating Therapy in Transfusional Iron Overload
Brief Title: Quantitative Susceptibility Mapping (QSM) to Guide Iron Chelating Therapy
Status: Recruiting | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Columbia University (Other); National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1706018263; R01DK116126-01A1 (NIH)
Record Dates: First submitted 2019-11-07; First posted 2019-11-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: MRI Scans
Keywords: Quantitative Susceptibility Mapping; Iron chelating therapy; Iron overload; Liver iron concentration; erythrocyte transfusion; liver transplantation; magnetic resonance imaging; thalassemia major
MeSH Terms: conditions — Iron Overload; beta-Thalassemia | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Liver explants to be obtained from the Department of Pathology and Cell Biology at Columbia after all clinical pathological examinations have been completed and the specimens would otherwise be discarded. Specimens are initially stored with identifying information but will be de-identified by the Study Pathologist prior to transport to Weill Cornell Medicine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with transfusional iron overload: The subject population of patients with transfusional iron overload awaiting liver transplant has been chosen because of the clinical indication for MRI examination every three months and the availability of liver explants for analysis after transplant. Explants will receive QSM or R2* MRI to provide a quantitative biophysical connection to liver iron concentration (LIC).
  Interventions: Radiation: Quantitative Susceptibility Mapping (QSM) Magnetic Resonance Imaging (MRI); Radiation: R2* Magnetic Resonance Imaging (MRI)
- Healthy subjects: Healthy control subjects over the age of 21 with no known hematological or liver disease and no contraindications for MRI
  Interventions: Radiation: Quantitative Susceptibility Mapping (QSM) Magnetic Resonance Imaging (MRI); Radiation: R2* Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Radiation: Quantitative Susceptibility Mapping (QSM) Magnetic Resonance Imaging (MRI) — Investigators will validate hepatic QSM (hQSM) using histological examination and chemical measurement of liver iron concentration (LIC). Patients will undergo clinical MRI in Aim 1. In patients with increased LIC their liver explants will undergo MRI, pathological examination, and chemical determination of the LIC.
Radiation: R2* Magnetic Resonance Imaging (MRI) — Investigators will be able to validate hQSM in measuring liver iron concentration (LIC) by comparing it to this traditional MRI technique

SUMMARY:
The overall goal of this research is to help develop a new magnetic resonance (MR) method, Quantitative Susceptibility Mapping (QSM), to improve the measurement of liver iron concentrations without the need for a liver biopsy. Measurement of liver iron is important to diagnose and treat patients who have too much iron in their bodies (iron overload). Liver iron measurements by current MRI methods (R2 and R2*) can be inaccurate because of the effects of fat, fibrosis and other abnormalities. QSM should not be affected by these factors and should be free of these errors. In this study, MRI measurements (QSM, R2 and R2*) of iron in patients before liver transplant will be compared with chemical analysis of iron in liver explants (livers removed from patients undergoing liver transplant). The liver explants would otherwise be discarded. Investigators expect that this study will show that the new MRI method, QSM, is superior to the current MRI methods, R2 and R2*.

DETAILED DESCRIPTION:
The overall objective of this research is to improve the safety of iron-chelating therapy (ICT) in patients with transfusional iron overload by developing an accurate non-invasive measurement of the liver iron concentration (LIC), the best measure of the body iron burden in all forms of systemic iron overload. The scientific premise is that quantitative susceptibility mapping (QSM) provides a quantitative biophysical connection to LIC. Safe ICT requires careful adjustment of the iron chelator dose to the body iron burden to optimize iron excretion while avoiding chelator toxicity, including gastrointestinal disorders, audiovisual impairment, neutropenia, arthropathy, growth retardation, and hepatic and renal failure. QSM enables accurate measurement of LIC by overcoming the inherent cellular interference in current R2 (=1/T2) and R2* (=R2+R2') estimates that lack a well-defined biophysical connection to the LIC. A fundamental biophysical limitation of the R2 and R2* approaches is that intravoxel contents other than iron, including fibrosis, steatosis and necroinflammation, also alter relaxation. In the liver, paramagnetic iron stored in ferritin and hemosiderin is the dominant susceptibility source for QSM. Consequently, magnetic susceptibility measured by QSM has a simple linear relationship with the concentration of iron in the liver and is little affected by fibrosis, steatosis and necroinflammation. The investigator's research plan has 3 specific aims:

Aim 1. Develop hQSM for accurate measurement of LIC without interfering errors. Investigators will optimize data acquisition and processing for free-breathing navigator acquisition with robust fat-water separation.

Aim 2. Validate hQSM using histology and chemical measurement of LIC in liver explants. Investigators will assess the accuracies of LICs measured by hQSM and R2* in patients before liver transplant with histologic examination using the reference standard of chemical measurement of LIC in liver explants.

Aim 3. Evaluate hQSM in patients with transfusional iron overload under ICT. In patients regularly transfused for thalassemia major, investigators will conduct a double-blind clinical study comparing the accuracy of hQSM and R2* in measuring annual changes in LIC, using regression against the year-long amount of iron administered in red blood cell transfusions and the year-long cumulative dose of iron chelator.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of thalassemia major
* Treatment with deferasirox formulated as Jadenu® as the sole iron chelating therapy (ICT)
* Regular transfusion with records maintained in the Cornell Thalassemia Program
* 2 years of age or older
* Females who are not pregnant

Inclusion Criteria (for healthy subjects):

* Men and women aged 21 years or older
* Able and willing to give consent
* No known hematological and liver disease
* No contraindications for MRI

Exclusion Criteria:

* A history of auditory or ocular toxicity related to ICT
* A history of poor adherence to prescribed therapy
* An inability to tolerate MRI examinations
* Treatment for mental illness
* Institutionalization or imprisonment

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy subjects will be selected from the community through personal contact and written description of the research, and online advertising.
  Subjects will be selected at Columbia from those awaiting liver transplant to be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Demonstration of efficacy of quantitative susceptibility mapping (QSM) MRI in quantifying liver iron concentration (LIC) | Five years
  Investigators will assess the accuracy of liver iron concentrations measured by QSM in patients before liver transplant with histologic examination using the gold standard chemical measurement of LIC in liver explants.

SECONDARY OUTCOMES:
Fibrosis as determined by in vivo R2*, an MRI method that provides quantitative information on iron levels | Five years
  R2* is an imaging method used in MRI. R2* = (1/T2*) where R2* is a relaxation rate measured in units of Hz ([1/sec]). R2* is commonly used to look at iron levels by measuring the relaxation times of hydrogen nuclei affected by iron. The presence of the iron results in the shortening of proton relaxation times (T2*), thus increasing R2*.
Fibrosis as determined by in vitro R2*, an MRI method that provides quantitative information on iron levels | Five years
  R2* is an imaging method used in MRI. R2* = (1/T2*) where R2* is a relaxation rate measured in units of Hz ([1/sec]). R2* is commonly used to look at iron levels by measuring the relaxation times of hydrogen nuclei affected by iron. The presence of the iron results in the shortening of proton relaxation times (T2*), thus increasing R2*.
Fibrosis as determined by in vivo hQSM, an MRI post-processing technique that provides quantitative information on iron levels | Five years
  Quantitative susceptibility mapping (QSM) is widely used by the imaging research community in applications to detect iron. Tissue can become magnetized in response to a magnetic field, and the extent of magnetization is known as susceptibility, which arises from unpaired electrons in iron or external sources such as contrast agents. QSM permits visualization of the sizes and shapes of iron sources, delivers precise estimates of iron concentrations (units: parts per billion [ppb] or parts per million [ppm]).
Fibrosis as determined by in vitro hQSM, an MRI post processing technique that provides quantitative information on iron levels | Five years
  Quantitative susceptibility mapping (QSM) is widely used by the imaging research community in applications to detect iron. Tissue can become magnetized in response to a magnetic field, and the extent of magnetization is known as susceptibility, which arises from unpaired electrons in iron or external sources such as contrast agents. QSM permits visualization of the sizes and shapes of iron sources, delivers precise estimates of iron concentrations (units: parts per billion [ppb] or parts per million [ppm]).
Steatosis as determined by in vivo R2*, an MRI method that provides quantitative information on iron levels | Five years
  R2* is an imaging method used in MRI. R2* = (1/T2*) where R2* is a relaxation rate measured in units of Hz ([1/sec]). R2* is commonly used to look at iron levels by measuring the relaxation times of hydrogen nuclei affected by iron. The presence of the iron results in the shortening of proton relaxation times (T2*), thus increasing R2*.
Steatosis as determined by in vitro R2*, an MRI method that provides quantitative information on iron levels | Five years
  R2* is an imaging method used in MRI. R2* = (1/T2*) where R2* is a relaxation rate measured in units of Hz ([1/sec]). R2* is commonly used to look at iron levels by measuring the relaxation times of hydrogen nuclei affected by iron. The presence of the iron results in the shortening of proton relaxation times (T2*), thus increasing R2*.
Steatosis as determined by in vivo hQSM, an MRI post-processing technique that provides quantitative information on iron levels | Five years
  Quantitative susceptibility mapping (QSM) is widely used by the imaging research community in applications to detect iron. Tissue can become magnetized in response to a magnetic field, and the extent of magnetization is known as susceptibility, which arises from unpaired electrons in iron or external sources such as contrast agents. QSM permits visualization of the sizes and shapes of iron sources, delivers precise estimates of iron concentrations (units: parts per billion [ppb] or parts per million [ppm]).
Steatosis as determined by in vitro hQSM, an MRI post-processing technique that provides quantitative information on iron levels | Five years
  Quantitative susceptibility mapping (QSM) is widely used by the imaging research community in applications to detect iron. Tissue can become magnetized in response to a magnetic field, and the extent of magnetization is known as susceptibility, which arises from unpaired electrons in iron or external sources such as contrast agents. QSM permits visualization of the sizes and shapes of iron sources, delivers precise estimates of iron concentrations (units: parts per billion [ppb] or parts per million [ppm]).
Necroinflammation as determined by in vivo R2*, an MRI method that provides quantitative information on iron levels | Five years
  R2* is an imaging method used in MRI. R2* = (1/T2*) where R2* is a relaxation rate measured in units of Hz ([1/sec]). R2* is commonly used to look at iron levels by measuring the relaxation times of hydrogen nuclei affected by iron. The presence of the iron results in the shortening of proton relaxation times (T2*), thus increasing R2*.
Necroinflammation as determined by in vitro R2*, an MRI method that provides quantitative information on iron levels | Five years
  R2* is an imaging method used in MRI. R2* = (1/T2*) where R2* is a relaxation rate measured in units of Hz ([1/sec]). R2* is commonly used to look at iron levels by measuring the relaxation times of hydrogen nuclei affected by iron. The presence of the iron results in the shortening of proton relaxation times (T2*), thus increasing R2*.
Necroinflammation as determined by in vivo hQSM, an MRI post-processing technique that provides quantitative information on iron levels | Five years
  Quantitative susceptibility mapping (QSM) is widely used by the imaging research community in applications to detect iron. Tissue can become magnetized in response to a magnetic field, and the extent of magnetization is known as susceptibility, which arises from unpaired electrons in iron or external sources such as contrast agents. QSM permits visualization of the sizes and shapes of iron sources, delivers precise estimates of iron concentrations (units: parts per billion [ppb] or parts per million [ppm]).
Necroinflammation as determined by in vitro hQSM, an MRI post-processing technique that provides quantitative information on iron levels | Five years
  Quantitative susceptibility mapping (QSM) is widely used by the imaging research community in applications to detect iron. Tissue can become magnetized in response to a magnetic field, and the extent of magnetization is known as susceptibility, which arises from unpaired electrons in iron or external sources such as contrast agents. QSM permits visualization of the sizes and shapes of iron sources, delivers precise estimates of iron concentrations (units: parts per billion [ppb] or parts per million [ppm]).

CONTACTS AND LOCATIONS:
Overall Officials: Gary M Brittenham, MD, Principal Investigator — Columbia University; Yi Wang, PhD, Principal Investigator — Weill Medical College of Cornell University; Sujit S Sheth, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Weill Cornell Medical College, New York, New York
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No